CLINICAL TRIAL: NCT02697526
Title: Influence of the Compression Method After Transradial Catheterization in Radial Artery
Brief Title: Differences in Radial Artery Occlusion From Two Different Compressive Methods Used in Patients in Order to Achieve Homeostasis After Transradial Catheterization and Their Repercussion in Artery Functionality and Hand Mobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: PR(AG)70/2006
Record Dates: First submitted 2016-02-23; First posted 2016-03-03 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-02

CONDITIONS: Transradial Catheterization
Keywords: radial artery; occlusion; functional; complications; consequences
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Terumo (Other): Patients in this arm will receive Terumo after catheterization
  Interventions: Other: Terumo
- Tensoplast (Other): Patients in this arm will receive Tensoplast after catheterization
  Interventions: Other: Tensoplast

INTERVENTIONS:
Other: Terumo
  Arms: Terumo
Other: Tensoplast
  Arms: Tensoplast

SUMMARY:
The aim of the study is to determine differences on radial artery occlusion from two compressive methods used after transradial catheterization and its functional impact on hand mobility.

DETAILED DESCRIPTION:
Changes in Allen's test and pulse oximetry will be evaluated at baseline, 1 week and 3 month of catheterization in both groups of patients in order to check the functionality of the communications between the ulnar and radial arteries. The repercussion of each compressive method on radial occlusion and artery revascularization will be assessed by eco-Doppler at any time. Changes in diameter of arterial lumen of radial and ulnar arteries as a consequence of radial occlusion will be done simultaneously of blood flow Doppler measurements. The possible impact of radial occlusion on hand mobility will be done using a dynamometer designed to evaluate strength (Endurance test) and muscular claudication (Rapid exchange test).

ELIGIBILITY:
Inclusion Criteria:

* Patients in whom at least the diagnostic catheterization has been done successfully by the radial artery route.
* Patients with a negative Allen's Clinical test showing hyperemia before 9 seconds after pressure release over the ulnar artery pulse.
* Patients showing a Barbeau pattern A,B or C with the pulsioximetric test after releasing pressure over the ulnar artery pulse.
* Patients that will be able to do the follow up visits at 1 week and 3 month.
* Signature of informed consent

Exclusion Criteria:

* Patients in that neither the diagnostic or therapeutic procedure has successfully done via the radial artery route.
* Patients with a positive Allen's test (no hyperemia) after pressure and release over the ulnar artery pulse.
* Patients showing a Barbeau pattern D with the pulsioximetric test after releasing pressure over the ulnar artery pulse.
* Inability to visit at 1 week and 3 month.
* Impossibility to obtain informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2007-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Determination of radial artery occlusion at baseline (before catheterization) | 1 day
  Determination of radial artery occlusion at baseline (before catheterization), 1 week and 3 month after angiography/angioplasty in both compressive methods
Determination of radial artery occlusion after catheterization | 1 week
  Determination of radial artery occlusion at baseline (before catheterization), 1 week and 3 month after angiography/angioplasty in both compressive methods
Determination of radial artery occlusion after catheterization | 3 month
  Determination of radial artery occlusion at baseline (before catheterization), 1 week and 3 month after angiography/angioplasty in both compressive methods

SECONDARY OUTCOMES:
Anatomic differences in radial and ulnar diameters | 3 month
  Anatomic differences in arterial lumen of radial and ulnar arteries (diameter)
Differences in radial and ulnar blood flow between compression methods | 3 month
  Differences in radial and ulnar blood flow as a consequence of radial occlusion
Differences in functional status at follow between compression groups | 1 day
  Differences in hand mobility at baseline, 1 week and 3 month of catheterization as a consequence of radial occlusion in relation with the compressive method used to achieve homeostasis.
Differences in functional status at follow between compression groups | 1 week
  Differences in hand mobility at baseline, 1 week and 3 month of catheterization as a consequence of radial occlusion in relation with the compressive method used to achieve homeostasis.
Differences in functional status at follow between compression groups | 3 month
  Differences in hand mobility at baseline, 1 week and 3 month of catheterization as a consequence of radial occlusion in relation with the compressive method used to achieve homeostasis.
Differences in functional status between occluded radial cohort and patent radial cohort | 1 day
  Differences in hand mobility at baseline, 1 week and 3 month in response to radial occlusion.
Differences in functional status between occluded radial cohort and patent radial cohort | 1 week
  Differences in hand mobility at baseline, 1 week and 3 month in response to radial occlusion.
Differences in functional status between occluded radial cohort and patent radial cohort | 3 month
  Differences in hand mobility at baseline, 1 week and 3 month in response to radial occlusion.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno García del Blanco, MD, PhD, Principal Investigator — Hospital Universitari Vall d'Hebron (Barcelona)
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Amoroso G, Kiemeneij F. Transradial access for primary percutaneous coronary intervention: the next standard of care? Heart. 2010 Sep;96(17):1341-4. doi: 10.1136/hrt.2010.196824. PMID 20801852
- [Background] Amoroso G, Laarman GJ, Kiemeneij F. Overview of the transradial approach in percutaneous coronary intervention. J Cardiovasc Med (Hagerstown). 2007 Apr;8(4):230-7. doi: 10.2459/01.JCM.0000263494.10865.0f. PMID 17413298
- [Background] Barbeau GR, Arsenault F, Dugas L, Simard S, Lariviere MM. Evaluation of the ulnopalmar arterial arches with pulse oximetry and plethysmography: comparison with the Allen's test in 1010 patients. Am Heart J. 2004 Mar;147(3):489-93. doi: 10.1016/j.ahj.2003.10.038. PMID 14999199
- [Background] Bassand JP. [Platelet antiaggregation treatment in the aftermath of GUSTO IV, TARGET, TACTICS, and CURE trials]. Rev Esp Cardiol. 2002 Jul;55(7):697-702. doi: 10.1016/s0300-8932(02)76686-4. Spanish. PMID 12113695
- [Background] Bassand JP, Afzal R, Eikelboom J, Wallentin L, Peters R, Budaj A, Fox KA, Joyner CD, Chrolavicius S, Granger CB, Mehta S, Yusuf S; OASIS 5 and OASIS 6 Investigators. Relationship between baseline haemoglobin and major bleeding complications in acute coronary syndromes. Eur Heart J. 2010 Jan;31(1):50-8. doi: 10.1093/eurheartj/ehp401. Epub 2009 Oct 12. PMID 19825809
- [Background] Biancari F, D'Andrea V, Di Marco C, Savino G, Tiozzo V, Catania A. Meta-analysis of randomized trials on the efficacy of vascular closure devices after diagnostic angiography and angioplasty. Am Heart J. 2010 Apr;159(4):518-31. doi: 10.1016/j.ahj.2009.12.027. PMID 20362708
- [Background] Brancati MF, Burzotta F, Coluccia V, Trani C. The occurrence of radial artery occlusion following catheterization. Expert Rev Cardiovasc Ther. 2012 Oct;10(10):1287-95. doi: 10.1586/erc.12.125. PMID 23190067
- [Background] Burstein JM, Gidrewicz D, Hutchison SJ, Holmes K, Jolly S, Cantor WJ. Impact of radial artery cannulation for coronary angiography and angioplasty on radial artery function. Am J Cardiol. 2007 Feb 15;99(4):457-9. doi: 10.1016/j.amjcard.2006.08.055. Epub 2006 Dec 20. PMID 17293183
- [Background] Campeau L. Percutaneous radial artery approach for coronary angiography. Cathet Cardiovasc Diagn. 1989 Jan;16(1):3-7. doi: 10.1002/ccd.1810160103. PMID 2912567
- [Background] Campeau L. Entry sites for coronary angiography and therapeutic interventions: from the proximal to the distal radial artery. Can J Cardiol. 2001 Mar;17(3):319-25. PMID 11264565
- [Background] Cardoso CO, Rodrigues LH, Cardoso CR, Yordi LM. Impact of radial artery cannulation on radial artery function. Am J Cardiol. 2007 Aug 15;100(4):743-4. doi: 10.1016/j.amjcard.2007.02.045. Epub 2007 May 25. No abstract available. PMID 17697842
- [Background] Cong X, Huang Z, Wu J, Wang J, Wen F, Fang L, Fan M, Liang C. Randomized Comparison of 3 Hemostasis Techniques After Transradial Coronary Intervention. J Cardiovasc Nurs. 2016 Sep-Oct;31(5):445-51. doi: 10.1097/JCN.0000000000000268. PMID 26002786
- [Background] Desai ND, Naylor CD, Kiss A, Cohen EA, Feder-Elituv R, Miwa S, Radhakrishnan S, Dubbin J, Schwartz L, Fremes SE; Radial Artery Patency Study Investigators. Impact of patient and target-vessel characteristics on arterial and venous bypass graft patency: insight from a randomized trial. Circulation. 2007 Feb 13;115(6):684-91. doi: 10.1161/CIRCULATIONAHA.105.567495. Epub 2007 Feb 5. PMID 17283268
- [Background] Dirksen MT, Ronner E, Laarman GJ, van Heerebeek L, Slagboom T, van der Wieken LR, van der Wouw PA, Kiemeneij F. Early discharge is feasible following primary percutaneous coronary intervention with transradial stent implantation under platelet glycoprotein IIb/IIIa receptor blockade. Results of the AGGRASTENT Trial. J Invasive Cardiol. 2005 Oct;17(10):512-7. PMID 16204742
- [Background] DOTTER CT, KRIPPAEHNE WW, JUDKINS MP. TRANSLUMINAL RECANALIZATION AND DILATATION IN ATHEROSCLEROTIC OBSTRUCTION OF FEMORAL POPLITEAL SYSTEM. Am Surg. 1965 Jul;31:453-9. No abstract available. PMID 14321155
- [Background] Dou K, Xu B, Yang Y, Chen J, Qiao S, Wang Y, Li J, Qin X, Yao M, Liu H, Wu Y, Chen J, Yuan J, You S, Gao R. Comparison of procedural and long-term outcomes between transradial and transfemoral approach in one-stage intervention for triple vessel coronary artery disease. J Interv Cardiol. 2014 Apr;27(2):108-16. doi: 10.1111/joic.12101. Epub 2014 Mar 4. PMID 24588842
- [Background] Elgharib NZ, Shah UH, Coppola JT. Transradial cardiac catheterization and percutaneous coronary intervention: a review. Coron Artery Dis. 2009 Dec;20(8):487-93. doi: 10.1097/MCA.0b013e32832f37fc. PMID 19641458
- [Background] Garcia del Blanco B, Hernandez Hernandez F, Rumoroso Cuevas JR, Trillo Nouche R. Spanish Cardiac Catheterization and Coronary Intervention Registry. 23rd official report of the Spanish Society of Cardiology Working Group on Cardiac Catheterization and Interventional Cardiology (1990-2013). Rev Esp Cardiol (Engl Ed). 2014 Dec;67(12):1013-23. doi: 10.1016/j.rec.2014.08.005. Epub 2014 Nov 11. PMID 25455754
- [Background] Gruntzig A. Transluminal dilatation of coronary-artery stenosis. Lancet. 1978 Feb 4;1(8058):263. doi: 10.1016/s0140-6736(78)90500-7. No abstract available. PMID 74678
- [Background] Gual-Capllonch F, García del Blanco B, Martí G, Batalla N, Domingo E, Ángel J. (2005). Diferències en les complicacions atribuïbles a l'accés radial entre el periode d'aprenentatge i el d'estabilització. Congrés Societat Catalana de Cardiologia- 2005
- [Background] Gual-Capllonch F, García del Blanco B, Martí G, Batalla N, Domingo E, Ángel J.(2004). Avaluació de la permeabilitat de l'artéria radial amb Doppler després de cateterisme via radial. Congrés Societat Catalana de Cardiologia-2004
- [Background] Gual-Capllonch F, García del Blanco B, Martí G, Otaegui I, Batalla N, Domingo E, Ángel J. (2005). Estudio con Doppler vascular de la permeabilidad de la arteria radial tras cateterismo cardiaco". Congreso Sociedad Española de Cardiología-2005.
- [Background] Heintzen MP, Schumacher T, Rath J, Ganschow U, Schoebel FC, Grabitz K, Vester EG, Leschke M, Kohler M, Strauer BE. [Incidence and therapy of peripheral arterial vascular complications after heart catheter examinations]. Z Kardiol. 1997 Apr;86(4):264-72. doi: 10.1007/s003920050058. German. PMID 9235798
- [Background] Hess CN, Peterson ED, Neely ML, Dai D, Hillegass WB, Krucoff MW, Kutcher MA, Messenger JC, Pancholy S, Piana RN, Rao SV. The learning curve for transradial percutaneous coronary intervention among operators in the United States: a study from the National Cardiovascular Data Registry. Circulation. 2014 Jun 3;129(22):2277-86. doi: 10.1161/CIRCULATIONAHA.113.006356. Epub 2014 Apr 22. PMID 24756064
- [Background] Koo BK, De Bruyne B. FFR in bifurcation stenting: what have we learned? EuroIntervention. 2010 Dec;6 Suppl J:J94-8. doi: 10.4244/EIJV6SUPJA15. PMID 21930499
- [Background] Jolly SS, Niemela K, Xavier D, Widimsky P, Budaj A, Valentin V, Lewis BS, Avezum A, Steg PG, Rao SV, Cairns J, Chrolavicius S, Yusuf S, Mehta SR. Design and rationale of the radial versus femoral access for coronary intervention (RIVAL) trial: a randomized comparison of radial versus femoral access for coronary angiography or intervention in patients with acute coronary syndromes. Am Heart J. 2011 Feb;161(2):254-260.e1-4. doi: 10.1016/j.ahj.2010.11.021. PMID 21315206
- [Background] Jolly SS, Yusuf S, Cairns J, Niemela K, Xavier D, Widimsky P, Budaj A, Niemela M, Valentin V, Lewis BS, Avezum A, Steg PG, Rao SV, Gao P, Afzal R, Joyner CD, Chrolavicius S, Mehta SR; RIVAL trial group. Radial versus femoral access for coronary angiography and intervention in patients with acute coronary syndromes (RIVAL): a randomised, parallel group, multicentre trial. Lancet. 2011 Apr 23;377(9775):1409-20. doi: 10.1016/S0140-6736(11)60404-2. Epub 2011 Apr 4. PMID 21470671
- [Background] Journal of Cardiovascular Nursing. (n.d.). Retrieved November 3, 2015, from http://journals.lww.com/jcnjournal/toc/publishahead
- [Background] Kamiya H, Ushijima T, Kanamori T, Ikeda C, Nakagaki C, Ueyama K, Watanabe G. Use of the radial artery graft after transradial catheterization: is it suitable as a bypass conduit? Ann Thorac Surg. 2003 Nov;76(5):1505-9. doi: 10.1016/s0003-4975(03)01018-x. PMID 14602276
- [Background] Kiemeneij F. Cost-effectiveness of transradial coronary access. J Invasive Cardiol. 2007 Aug;19(8):354. No abstract available. PMID 17712205
- [Background] Kiemeneij F, Laarman GJ. Percutaneous transradial artery approach for coronary stent implantation. Cathet Cardiovasc Diagn. 1993 Oct;30(2):173-8. doi: 10.1002/ccd.1810300220. PMID 8221875
- [Background] Kiemeneij F, Laarman GJ, Odekerken D, Slagboom T, van der Wieken R. A randomized comparison of percutaneous transluminal coronary angioplasty by the radial, brachial and femoral approaches: the access study. J Am Coll Cardiol. 1997 May;29(6):1269-75. doi: 10.1016/s0735-1097(97)00064-8. PMID 9137223
- [Background] Kiemeneij F, Vajifdar BU, Eccleshall SC, Laarman G, Slagboom T, van der Wieken R. Measurement of radial artery spasm using an automatic pullback device. Catheter Cardiovasc Interv. 2001 Dec;54(4):437-41. doi: 10.1002/ccd.1307. PMID 11747176
- [Background] Kiviniemi T, Airaksinen KE, Rubboli A, Biancari F, Valencia J, Lip GY, Karjalainen PP, Weber M, Laine M, Kirchhof P, Schlitt A; AFCAS (Management of patients with Atrial Fibrillation undergoing Coronary Artery Stenting) study group. Bridging therapy with low molecular weight heparin in patients with atrial fibrillation undergoing percutaneous coronary intervention with stent implantation: the AFCAS study. Int J Cardiol. 2015 Mar 15;183:105-10. doi: 10.1016/j.ijcard.2015.01.056. Epub 2015 Jan 27. PMID 25662060
- [Background] Klinke WP, Hilton JD, Warburton RN, Warburton WP, Tan RP. Comparison of treatment outcomes in patients > or =80 years undergoing transradial versus transfemoral coronary intervention. Am J Cardiol. 2004 May 15;93(10):1282-5. doi: 10.1016/j.amjcard.2004.02.015. PMID 15135705
- [Background] Kurisu S, Mitsuba N, Kato Y, Ishibashi K, Dohi Y, Nishioka K, Kihara Y. External side-compression of radial artery: a simple technique for successful advancement of guidewires through the radial approach. J Interv Cardiol. 2011 Oct;24(5):397-400. doi: 10.1111/j.1540-8183.2011.00668.x. Epub 2011 Aug 25. PMID 21883471
- [Background] Kusztal M, Weyde W, Letachowicz K, Golebiowski T, Letachowicz W. Anatomical vascular variations and practical implications for access creation on the upper limb. J Vasc Access. 2014;15 Suppl 7:S70-5. doi: 10.5301/jva.5000257. Epub 2014 Apr 17. PMID 24817459
- [Background] Lewis BS, Mehta SR, Fox KA, Halon DA, Zhao F, Peters RJ, Keltai M, Budaj A, Yusuf S; CURE trial investigators. Benefit of clopidogrel according to timing of percutaneous coronary intervention in patients with acute coronary syndromes: further results from the Clopidogrel in Unstable angina to prevent Recurrent Events (CURE) study. Am Heart J. 2005 Dec;150(6):1177-84. doi: 10.1016/j.ahj.2005.01.044. PMID 16338255
- [Background] Louvard Y, Lefevre T, Allain A, Morice M. Coronary angiography through the radial or the femoral approach: The CARAFE study. Catheter Cardiovasc Interv. 2001 Feb;52(2):181-7. doi: 10.1002/1522-726x(200102)52:23.0.co;2-g. PMID 11170325
- [Background] Martí Aguasa G., Otaegui Irurueta I., García del Blanco B., Alguersuari Cabiscol J., Ayats M., Domingo Ribas E., Angel Ferrer J., Anivarro Blanco I., Soler Soler J. (2006). Evolució a mig termini de l'oclusió arterial radial després del cateterisme cardiac. Congrés de la Societat Caltalana de Cardiologia-2006
- [Background] Madssen E, Haere P, Wiseth R. Radial artery diameter and vasodilatory properties after transradial coronary angiography. Ann Thorac Surg. 2006 Nov;82(5):1698-702. doi: 10.1016/j.athoracsur.2006.06.017. PMID 17062231
- [Background] Mohite PN, Thingnam SK, Saxena AK. Radial artery compression in incomplete palmar arch for radial artery harvesting. Asian Cardiovasc Thorac Ann. 2014 May;22(4):416-20. doi: 10.1177/0218492313490936. Epub 2013 Oct 16. PMID 24771729
- [Background] Morice MC, Serruys PW, Sousa JE, Fajadet J, Ban Hayashi E, Perin M, Colombo A, Schuler G, Barragan P, Guagliumi G, Molnar F, Falotico R; RAVEL Study Group. Randomized Study with the Sirolimus-Coated Bx Velocity Balloon-Expandable Stent in the Treatment of Patients with de Novo Native Coronary Artery Lesions. A randomized comparison of a sirolimus-eluting stent with a standard stent for coronary revascularization. N Engl J Med. 2002 Jun 6;346(23):1773-80. doi: 10.1056/NEJMoa012843. PMID 12050336
- [Background] Nagai S, Abe S, Sato T, Hozawa K, Yuki K, Hanashima K, Tomoike H. Ultrasonic assessment of vascular complications in coronary angiography and angioplasty after transradial approach. Am J Cardiol. 1999 Jan 15;83(2):180-6. doi: 10.1016/s0002-9149(98)00821-2. PMID 10073818
- [Background] Nikolsky E, Mehran R, Halkin A, Aymong ED, Mintz GS, Lasic Z, Negoita M, Fahy M, Krieger S, Moussa I, Moses JW, Stone GW, Leon MB, Pocock SJ, Dangas G. Vascular complications associated with arteriotomy closure devices in patients undergoing percutaneous coronary procedures: a meta-analysis. J Am Coll Cardiol. 2004 Sep 15;44(6):1200-9. doi: 10.1016/j.jacc.2004.06.048. PMID 15364320
- [Background] Pancholy SB, Joshi P, Shah S, Rao SV, Bertrand OF, Patel TM. Effect of Vascular Access Site Choice on Radiation Exposure During Coronary Angiography: The REVERE Trial (Randomized Evaluation of Vascular Entry Site and Radiation Exposure). JACC Cardiovasc Interv. 2015 Aug 17;8(9):1189-1196. doi: 10.1016/j.jcin.2015.03.026. Epub 2015 Jul 22. PMID 26210808
- [Background] Pancholy S, Coppola J, Patel T, Roke-Thomas M. Prevention of radial artery occlusion-patent hemostasis evaluation trial (PROPHET study): a randomized comparison of traditional versus patency documented hemostasis after transradial catheterization. Catheter Cardiovasc Interv. 2008 Sep 1;72(3):335-340. doi: 10.1002/ccd.21639. PMID 18726956
- [Background] Pandie S, Mehta SR, Cantor WJ, Cheema AN, Gao P, Madan M, Niemela K, Rao SV, Schwalm JD, Valentin V, Velianou JL, Jolly SS. Radial Versus Femoral Access for Coronary Angiography/Intervention in Women With Acute Coronary Syndromes: Insights From the RIVAL Trial (Radial Vs femorAL access for coronary intervention). JACC Cardiovasc Interv. 2015 Apr 20;8(4):505-12. doi: 10.1016/j.jcin.2014.11.017. PMID 25907080
- [Background] Pedreros, P., Lamich, R., Aguirre, A., Romero, C., Chamorro, H., & Donoso, M. (2010). Evaluación a largo plazo del impacto funcional y estructural de la arteria radial post acceso en intervencionismo coronario. Revista Chilena de Cardiología, 29(2), 193-198.
- [Background] Philippe F, Larrazet F, Meziane T, Dibie A. Comparison of transradial vs. transfemoral approach in the treatment of acute myocardial infarction with primary angioplasty and abciximab. Catheter Cardiovasc Interv. 2004 Jan;61(1):67-73. doi: 10.1002/ccd.10675. PMID 14696162
- [Background] Pillay D, Lam KH, Muda MN, Hamid Z. Transradial coronary angioplasty and stenting--immediate results and 3-month clinical follow-up in the first 50 patients performed at the National Heart Institute. Med J Malaysia. 2000 Dec;55(4):467-72. PMID 11221159
- [Background] Politi L, Aprile A, Paganelli C, Amato A, Zoccai GB, Sgura F, Monopoli D, Rossi R, Modena MG, Sangiorgi GM. Randomized clinical trial on short-time compression with Kaolin-filled pad: a new strategy to avoid early bleeding and subacute radial artery occlusion after percutaneous coronary intervention. J Interv Cardiol. 2011 Feb;24(1):65-72. doi: 10.1111/j.1540-8183.2010.00584.x. Epub 2010 Aug 29. PMID 20807305
- [Background] Ratib K, Chong AY, Routledge H, Nolan J. Spasm and occlusion in contemporary radial practice. JACC Cardiovasc Interv. 2010 Aug;3(8):885-6; author reply 886-7. doi: 10.1016/j.jcin.2010.06.008. No abstract available. PMID 20723865
- [Background] Rechenmacher SJ, Fang JC. Bridging Anticoagulation: Primum Non Nocere. J Am Coll Cardiol. 2015 Sep 22;66(12):1392-403. doi: 10.1016/j.jacc.2015.08.002. PMID 26383727
- [Background] Rubboli A, Colletta M, Valencia J, Capecchi A, Franco N, Zanolla L, La Vecchia L, Piovaccari G, Di Pasquale G; WARfarin and Coronary STENTing (WAR-STENT) Study Group. Periprocedural management and in-hospital outcome of patients with indication for oral anticoagulation undergoing coronary artery stenting. J Interv Cardiol. 2009 Aug;22(4):390-7. doi: 10.1111/j.1540-8183.2009.00468.x. Epub 2009 May 6. PMID 19453820
- [Background] Sabate M, Cequier A, Iniguez A, Serra A, Hernandez-Antolin R, Mainar V, Valgimigli M, Tespili M, den Heijer P, Bethencourt A, Vazquez N, Gomez-Hospital JA, Baz JA, Martin-Yuste V, van Geuns RJ, Alfonso F, Bordes P, Tebaldi M, Masotti M, Silvestro A, Backx B, Brugaletta S, van Es GA, Serruys PW. Everolimus-eluting stent versus bare-metal stent in ST-segment elevation myocardial infarction (EXAMINATION): 1 year results of a randomised controlled trial. Lancet. 2012 Oct 27;380(9852):1482-90. doi: 10.1016/S0140-6736(12)61223-9. Epub 2012 Sep 3. PMID 22951305
- [Background] Saito S, Ikei H, Hosokawa G, Tanaka S. Influence of the ratio between radial artery inner diameter and sheath outer diameter on radial artery flow after transradial coronary intervention. Catheter Cardiovasc Interv. 1999 Feb;46(2):173-8. doi: 10.1002/(SICI)1522-726X(199902)46:23.0.CO;2-4. PMID 10348538
- [Background] Sanmartin M, Goicolea J, Ocaranza R, Cuevas D, Calvo F. Vasoreactivity of the radial artery after transradial catheterization. J Invasive Cardiol. 2004 Nov;16(11):635-8. PMID 15550733
- [Background] Santas E, Bodi V, Sanchis J, Nunez J, Mainar L, Minana G, Chorro FJ, Llacer A. The left radial approach in daily practice. A randomized study comparing femoral and right and left radial approaches. Rev Esp Cardiol. 2009 May;62(5):482-90. doi: 10.1016/s1885-5857(09)71830-4. English, Spanish. PMID 19406062
- [Background] Serruys PW, Chevalier B, Dudek D, Cequier A, Carrie D, Iniguez A, Dominici M, van der Schaaf RJ, Haude M, Wasungu L, Veldhof S, Peng L, Staehr P, Grundeken MJ, Ishibashi Y, Garcia-Garcia HM, Onuma Y. A bioresorbable everolimus-eluting scaffold versus a metallic everolimus-eluting stent for ischaemic heart disease caused by de-novo native coronary artery lesions (ABSORB II): an interim 1-year analysis of clinical and procedural secondary outcomes from a randomised controlled trial. Lancet. 2015 Jan 3;385(9962):43-54. doi: 10.1016/S0140-6736(14)61455-0. Epub 2014 Sep 14. PMID 25230593
- [Background] Serruys PW, de Jaegere P, Kiemeneij F, Macaya C, Rutsch W, Heyndrickx G, Emanuelsson H, Marco J, Legrand V, Materne P, et al. A comparison of balloon-expandable-stent implantation with balloon angioplasty in patients with coronary artery disease. Benestent Study Group. N Engl J Med. 1994 Aug 25;331(8):489-95. doi: 10.1056/NEJM199408253310801. PMID 8041413
- [Background] Stefanini GG, Byrne RA, Serruys PW, de Waha A, Meier B, Massberg S, Juni P, Schomig A, Windecker S, Kastrati A. Biodegradable polymer drug-eluting stents reduce the risk of stent thrombosis at 4 years in patients undergoing percutaneous coronary intervention: a pooled analysis of individual patient data from the ISAR-TEST 3, ISAR-TEST 4, and LEADERS randomized trials. Eur Heart J. 2012 May;33(10):1214-22. doi: 10.1093/eurheartj/ehs086. Epub 2012 Mar 24. PMID 22447805
- [Background] Stella PR, Kiemeneij F, Laarman GJ, Odekerken D, Slagboom T, van der Wieken R. Incidence and outcome of radial artery occlusion following transradial artery coronary angioplasty. Cathet Cardiovasc Diagn. 1997 Feb;40(2):156-8. doi: 10.1002/(sici)1097-0304(199702)40:23.0.co;2-a. PMID 9047055
- [Background] Urban P, Meredith IT, Abizaid A, Pocock SJ, Carrie D, Naber C, Lipiecki J, Richardt G, Iniguez A, Brunel P, Valdes-Chavarri M, Garot P, Talwar S, Berland J, Abdellaoui M, Eberli F, Oldroyd K, Zambahari R, Gregson J, Greene S, Stoll HP, Morice MC; LEADERS FREE Investigators. Polymer-free Drug-Coated Coronary Stents in Patients at High Bleeding Risk. N Engl J Med. 2015 Nov 19;373(21):2038-47. doi: 10.1056/NEJMoa1503943. Epub 2015 Oct 14. PMID 26466021
- [Background] Valsecchi O, Vassileva A, Musumeci G, Rossini R, Tespili M, Guagliumi G, Mihalcsik L, Gavazzi A, Ferrazzi P. Failure of transradial approach during coronary interventions: anatomic considerations. Catheter Cardiovasc Interv. 2006 Jun;67(6):870-8. doi: 10.1002/ccd.20732. PMID 16649233